CLINICAL TRIAL: NCT02246556
Title: Dichoptic Virtual Reality Therapy for Amblyopia in Adults
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Recruitment inadequate and investigators leaving the study institution for new positions.
Sponsor: University of California, San Francisco (Other)
Responsible Party: Principal Investigator, Marc Levin, Assistant Professor, Neuro-ophthalmology, University of California, San Francisco
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 14-14212; 093955 (Other: UCSF)
Record Dates: First submitted 2014-09-17; First posted 2014-09-22 (Estimated); Last update posted 2017-05-03 (Actual); Status verified 2017-05

CONDITIONS: Amblyopia; Anisometropia; Strabismus
Keywords: Amblyopia; Dichoptic; Virtual reality; Stereopsis; Stereo vision; Visual acuity; Binocular
MeSH Terms: conditions — Amblyopia; Anisometropia; Strabismus | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Patching therapy (Active Comparator): Patching treatment followed by crossover to dichoptic virtual reality video game treatment arm using Diplopia (TM) software developed for the Oculus Rift (R) game system.
  Interventions: Other: Patching therapy
- Dioptic (non-dichoptic) therapy (Active Comparator): Dioptic (non-dichoptic) therapy followed by crossover to dichoptic virtual reality video game treatment arm using Diplopia (TM) software developed for the Oculus Rift (R) game system.
  Interventions: Device: Dioptic (non-dichoptic) therapy
- Dichoptic therapy (Experimental): Dichoptic virtual reality video game treatment using Diplopia (TM) software developed for the Oculus Rift (R) game system.
  Interventions: Device: Dichoptic therapy

INTERVENTIONS:
Device: Dichoptic therapy — Dichoptic virtual reality video game therapy with Diplopoia (TM) software developed for the Oculus Rift (R) gaming system
  Arms: Dichoptic therapy
Other: Patching therapy — Conventional patching therapy followed by crossover to the dichoptic virtual reality video game therapy with Diplopia (TM) software
  Arms: Patching therapy
Device: Dioptic (non-dichoptic) therapy — Dioptic (non-dichoptic) video game therapy followed by crossover to the dichoptic virtual reality video game therapy with Diplopia (TM) software
  Arms: Dioptic (non-dichoptic) therapy

SUMMARY:
This was a randomized, masked, controlled study of the effect of a virtual reality, binocular, 3-dimensional video game on visual acuity and stereopsis in adult patients with amblyopia. The trial has been halted as of June 2016 and will not be evaluating any new subjects for enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Interpupillary distance of 60-66 mm
* Age 15-40
* Anisometropic amblyopia or strabismic amblyopia
* Best corrected visual acuity of 20/30 or worse in the amblyopic eye
* No prior therapeutic use of the software
* No other ongoing therapies including patching or recent eye muscle surgery
* No vested interest in the product
* Ability attend visits and complete the training session, and to stop the intervention after the specified intervention period

Exclusion Criteria:

* Stimulus-deprivation amblyopia.
* Organic lesions of the eye preventing the establishment of good vision (eg. media opacities, abnormalities in the fundus or optic nerve).
* Lesions of the brain preventing the establishment of good vision (eg. cortical visual impairment).
* Establishment of normal vision by refractive adaptation (wearing glasses after presentation).
* Patients diagnosed with Photosensitive Epilepsy.
* Inability to comply with the follow-up visits required.
* History of pathologic nystagmus (congenital or sensory).

Ages: 15 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 17 (Actual)
Dates: Start 2014-10; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Change in visual acuity | 3 weeks, 6 weeks, and 6 months

SECONDARY OUTCOMES:
Change in stereopsis | 3 weeks, 6 weeks, and 6 months
Quality of life | 3 weeks, 6 weeks, and 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- University of California, San Francisco, San Francisco, California, United States